CLINICAL TRIAL: NCT03647969
Title: Modified FOLFOX Plus/Minus Nivolumab and Ipilimumab vs. FLOT Plus Nivolumab in Patients With Previously Untreated Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction - A Randomized Phase 2 Trial.
Brief Title: Modified FOLFOX Plus/Minus Nivolumab and Ipilimumab vs. FLOT Plus Nivolumab in Patients With Previously Untreated Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-STO-0417; 2017-002080-18 (EudraCT Number); CA209-9KG (Other Grant/Funding Number: Bristol Myers-Squibb)
Record Dates: First submitted 2018-06-28; First posted 2018-08-27 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Adenocarcinoma of the Stomach; GastroEsophageal Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mFOLFOX/Nivolumab/Ipilimumab A/A1 (Experimental): Nivolumab 240mg "Flatdose" i.v. d1 over 30 min every 2 weeks followed by Ipilimumab 1mg/kg i.v. d1 over 30 min every 6 weeks followed by FOLFOX Oxaliplatin 85 mg/m² iv 2hrs (day 1), Leucovorin 400 mg/m2 iv 2hrs (day 1), Fluorouracil 400 mg/m² iv bolus (day 1), and Fluorouracil 2400 mg/m² iv continuous infusion over 44 hours (day 1+2) every 2 weeks until disease progression or inacceptable toxicity or end of study treatment.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: mFOLFOX
- mFOLFOX/Nivolumab/Ipilimumab sequential A2 (Experimental): 3 cycles of induction chemotherapy with FOLFOX: FOLFOX Oxaliplatin 85 mg/m² iv 2hrs (day 1), Leucovorin 400 mg/m2 iv 2hrs (day 1), Fluorouracil 400 mg/m² iv bolus (day 1), and Fluorouracil 2400 mg/m² iv continuous infusion over 44 hours (day 1+2) every 2 weeks followed by immunotherapy consisting of: 4 administrations of Nivolumab 240mg "Flatdose" i.v. d1 over 30 minutes every 2 weeks and 2 administrations of Ipilimumab 1mg/kg i.v. d1 over 30 minutes every 6 weeks
  Sequence as described may be repeated starting two weeks after last administration of immunotherapy once, or, if medically reasonable, for an unlimited number of repetitions upon investigator decision. After discontinuation of chemotherapy, immunotherapy will be continued consisting of:
  Nivolumab at 240mg "Flatdose" i.v. d1 every 2 weeks and Ipilimumab at 1mg/kg i.v. d1 every 6 weeks until disease progression or inacceptable toxicity or end of study treatment.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: mFOLFOX
- mFOLFOX B (Active Comparator): FOLFOX Oxaliplatin 85 mg/m² iv 2hrs (day 1), Leucovorin 400 mg/m2 iv 2hrs (day 1), Fluorouracil 400 mg/m² iv bolus (day 1), and Fluorouracil 2400 mg/m² iv continuous infusion over 44 hours (day 1+2) every 2 weeks until disease progression or inacceptable toxicity or end of study treatment.
  Interventions: Drug: mFOLFOX
- FLOT/Nivolumab C (Experimental): Nivolumab 240mg "Flatdose" i.v. d1 every 2 weeks followed by FLOT: Docetaxel 50mg/², Oxaliplatin 85 mg/m², leucovorin 200 mg/m² on day 1 and fluorouracil 2600 mg/m² IV continuous infusion over 24 hours every 2 weeks until disease progression or inacceptable toxicity or end of study treatment. After completion or discontinuation of chemotherapy, immunotherapy may be continued consisting of: Nivolumab at 240mg "Flatdose" i.v. d1 every 2 weeks Chemotherapy can also be administered per local standard.
  Interventions: Drug: Nivolumab; Drug: FLOT

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240mg "Flatdose" i.v. d1 over 30 minutes every 2 weeks
  Arms: FLOT/Nivolumab C; mFOLFOX/Nivolumab/Ipilimumab A/A1; mFOLFOX/Nivolumab/Ipilimumab sequential A2
Drug: Ipilimumab — 1mg/kg i.v. d1 over 30 minutes every 6 weeks
  Arms: mFOLFOX/Nivolumab/Ipilimumab A/A1; mFOLFOX/Nivolumab/Ipilimumab sequential A2
Drug: mFOLFOX — Oxaliplatin at a dose of 85 mg/m² iv over two hours (day 1), Leucovorin at a dose of 400 mg/m2 iv over two hours (day 1), Fluorouracil at a dose of 400 mg/m² iv bolus (day 1), and Fluorouracil at a dose of 2400 mg/m² iv continuous infusion over 44 hours (day 1+2) every 2 weeks
  Arms: mFOLFOX B; mFOLFOX/Nivolumab/Ipilimumab A/A1; mFOLFOX/Nivolumab/Ipilimumab sequential A2
Drug: FLOT — Docetaxel at a dose of 50 mg/m² iv over one hour (day 1), Oxaliplatin at a dose of 85 mg/m² iv over two hours (day 1), Leucovorin* at a dose of 200 mg/m² iv over one hour (day 1), Fluorouracil at a dose of 2600 mg/m² iv over 24 hours (day 1) every 2 weeks
  * Note: Leucovorin can be replaced by sodium folinate that is given according to local guideline.
  Arms: FLOT/Nivolumab C

SUMMARY:
Patients with Her2 negative, previously untreated metastatic esophagogastric adenocarcinoma will be treated with modified FOLFOX, with modified FOLFOX plus Nivolumab and Ipilimumab or FLOT plus Nivolumab. The groups will be compared for time until progression of the disease (primary endpoint) as well as for response to the treatment, overall survival, safety/tolerability of the treatment and quality of life.

DETAILED DESCRIPTION:
This is a randomized, open labelled multicenter phase II trial, followed by a non-randomized arm.

Patients with Her2 negative, previously untreated metastatic esophagogastric adenocarcinoma will be randomized to receive either modified FOLFOX (Oxaliplatin at a dose of 85 mg/m² iv over two hours (day 1), Leucovorin at a dose of 400 mg/m2 iv over two hours (day 1), Fluorouracil at a dose of 400 mg/m² iv bolus (day 1), and Fluorouracil at a dose of 2400 mg/m² iv continuous infusion over 44 hours (day 1+2), every 2 weeks) alone, modified FOLFOX plus Nivolumab (240mg "Flatdose" i.v. d1 every 2 weeks) and Ipilimumab (1mg/kg i.v. d1 every 6 weeks) or sequential treatment (three cycles of induction chemotherapy with modified FOLFOX followed by immunotherapy consisting of 4 administrations of Nivolumab at 240mg "Flatdose" i.v. d1 every 2 weeks and 2 administrations of Ipilimumab at 1mg/kg i.v. d1 every 6 weeks, this sequence may be repeated starting two weeks after last administration of immunotherapy once, or, if medically reasonable, for an unlimited number of repetitions upon investigator decision; after completion or discontinuation of chemotherapy, immunotherapy will be continued consisting of Nivolumab at 240mg "Flatdose" i.v. d1 every 2 weeks and Ipilimumab at 1mg/kg i.v. d1 every 6 weeks). In a non-randomized arm, patients receive Nivolumab 240mg "Flatdose" i.v. d1 every 2 weeks and FLOT (Docetaxel 50mg/², Oxaliplatin 85 mg/m², leucovorin 200 mg/m² on day 1 and fluorouracil 2600 mg/m² IV continuous infusion over 24 hours) every 2 weeks. After completion or discontinuation of chemotherapy, immunotherapy may be continued (Nivolumab at 240mg "Flatdose" i.v. d1 every 2 weeks).

Treatment in every arm will be given for a maximum of 24 months or until disease progression or inacceptable toxicity or end of study treatment.

The primary objective is to determine the clinical performance of the experimental regimen in patients with previously untreated HER2 negative locally advanced or metastatic esophagogastric adenocarcinoma in terms of progression free survival (acc. to RECIST v1.1).

Secondary objectives are to determine efficacy in terms of objective response rate (acc. to RECIST v1.1) and overall survival, as well as tolerability (acc. to NCI CTC AE v4.03) of the experimental regimen. In addition histopathological types and molecular parameters such as immune cell composition and PD-L1 expression as determined by quantitative mRNA (RT-PCR) will be correlated with efficacy in an exploratory analysis.

257 subjects (59 in the control arm, 89 in the experimental treatment group A1, 59 in the experimental treatment group A2 and 50 in the experimental treatment group C) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must have inoperable, advanced or metastatic GC or GEJ adenocarcinoma.
2. Subjects must have HER2-negative disease defined as either IHC 0 or I+ or IHC 2+, the latter in combination with ISH-, as assessed locally on a primary or metastatic tumour.
3. Subject must be previously untreated with systemic treatment given as primary therapy for advanced or metastatic disease.
4. Prior adjuvant or neoadjuvant chemotherapy, radiotherapy and/or chemoradiotherapy are permitted as long as the last administration of the last regimen (whichever was given last) occurred at least 6 months prior to randomization/enrolment.
5. Palliative radiotherapy is allowed and must be completed 2 weeks prior to randomization/enrolment.
6. Subjects must have measurable or evaluable non-measurable disease as assessed by the investigator, according to RECIST v1.1 (Appendix D).
7. ECOG performance status score of 0 or 1 (Appendix B).
8. Life expectancy > 12 weeks
9. Screening laboratory values must meet the following criteria (using NCI CTCAE v.4.03):

   1. WBC ≥ 2000/uL
   2. Neutrophils ≥ 1500/µL
   3. Platelets ≥ 100x10^3/µL
   4. Hemoglobin ≥ 9.0 g/dL
   5. Serum creatinine ≤ 1.5 x ULN
   6. AST ≤ 3.0 x ULN (or ≤ 5.0X ULN if liver metastates are present)
   7. ALT ≤ 3.0 x ULN (or ≤ 5.0X ULN if liver metastates are present)
   8. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome who must have a total bilirubin level of < 3.0 x ULN)
10. Males and Females* ≥ 18 years of age

    *There are no data that indicate special gender distribution. Therefore patients will be enrolled in the study gender-independently.
11. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care.
12. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
13. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug. Women must not be breastfeeding.
14. WOCBP must agree to follow instructions for method(s) of contraception for a period of 30 days (duration of ovulatory cycle) plus the time required for the investigational drug to undergo 5 half-lives. The terminal half-lives of nivolumab and ipilimumab are approximately 25 days and 15 days, respectively. WOCBP should use an adequate method to avoid pregnancy for approximately 5 months (30 days plus the time required for nivolumab to undergo 5 half-lives) after the last dose of investigational drug.
15. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for a period of 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo 5 half-lives. The terminal half-lives of nivolumab and ipilimumab are approximately 25 days and 15 days, respectively. Males who are sexually active with WOCBP must continue contraception for approximately 7 months (90 days plus the time required for nivolumab to undergo 5 half-lives) after the last dose of investigational drug. In addition, male subjects must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

1. Malignancies other than disease under study within 5 years prior to inclusion, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
2. Subjects with untreated symptomatic CNS metastases. Subjects are eligible if CNS metastases are asymptomatic (this includes patients with unknown CNS metastatic status who have no clinical signs of CNS metastases) or those with asymptomatic or symptomatic CNS who are adequately treated and are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to randomization/enrolment. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of < 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to randomization/enrolment. Patients with unknown CNS metastatic status and any clinical signs indicative of CNS metastases are eligible if CNS metastases are excluded using CT and/or MRI scans, or CNS metastases are confirmed but adequately treated as described above.
3. Subjects with active, known, or suspected autoimmune disease. Subjects with Type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. For any cases of uncertainty, it is recommended that the medical monitor be consulted prior to signing informed consent.
4. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
5. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
6. All toxicities attributed to prior anti-cancer therapy other than hearing loss, alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 4.03) or baseline before administration of study drug.
7. > Grade 1 peripheral neuropathy according to CTCAE version 4.0
8. Known Dihydropyrimidine dehydrogenase (DPD) deficiency
9. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive study drug.
10. Ascites which cannot be controlled with appropriate interventions.
11. Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry; congestive heart failure NYHA grade 3 and 4
12. Significant acute or chronic infections including, among others:

    1. Positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
    2. Any positive test result for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
13. History of allergy or hypersensitivity to study drugs or any constituent of the products
14. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
15. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) Arm A and B | Up to 3 years
  PFS, defined as time from randomization to the date of first observed disease progression as assessed by the investigator using CT criteria or death from any cause assessed every 8 weeks for up to 3 years Arm A versus Arm B
Progression-free Survival rate at 6 months Arm A2 and C | 6 months after randomization/enrolment
  PFS rate at 6 months is defined as proportion of patients being known to be alive and free of disease progression as assessed by the investigator using CT criteria at 6 months after randomization/enrolment

SECONDARY OUTCOMES:
Progression-free survival (PFS) Arm A1, A2, C | Up to 3 years
  PFS, defined as time from randomization/enrolment to the date of first observed disease progression as assessed by the investigator using CT criteria or death from any cause assessed every 8 weeks for up to 3 years for Arm A1, Arm A2 and Arm C
Progression-free Survival rate at 6 months Arms A and B | 6 months after randomization
  PFS rate at 6 months is defined as proportion of patients being known to be alive and free of disease progression as assessed by the investigator using CT criteria at 6 months after randomization
Overall Response Rate (ORR) | Up to 2 years
  ORR defined as proportion of patients with complete or partial response (CR + PR) as assessed according to RECIST criteria every 8 weeks for up to 2 years
Duration of response and disease stabilization | Up to 3 years
  Duration of response and disease stabilization defined as time from documentation of tumor response (CR, PR) or disease stabilization (SD) according to RECIST criteria to disease progression or death for up to 3 years
Overall survival (OS) | Up to 3 years
  Overall survival according to Kaplan-Meier assessed from randomization/enrolment to the date of death from any cause
Incidence and severity of adverse events | Up to 27 months
  incidence and severity of adverse events according to CTCAE (Common Terminology Criteria for Adverse Events) Version 4.03 criteria as assessed every 2 weeks during treatment and until 100 days after the last dose of study drug
Patient reported outcomes: Quality of life | Up to 3 years
  Quality of life as measured by questionnaire EORTC-QLQ-C30 from randomization every 8 weeks until EOT and afterwards every 3 months until first observed disease progression or death for up to 3 years
Progression-free survival (PFS) by PD-L1 expression status | Up to 3 years
  Subgroup analysis of PFS, defined as time from randomization/enrolment to the date of first observed disease progression as assessed by the investigator using CT criteria or death from any cause assessed every 8 weeks for up to 3 years, according to PD-L1 expression status
Overall survival (OS) by PD-L1 expression status | Up to 3 years
  Subgroup analysis of overall survival according to Kaplan-Meier assessed from randomization/enrolment to the date of death from any cause according to PD-L1 expression status

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Chair — Krankenhaus Nordwest
Locations (27):
- Germany (27):
  - Klinikum St. Marien Amberg, Amberg
  - Klinikum Aschaffenburg, Aschaffenburg
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Charité CVK, Berlin
  - HELIOS Klinikum Berlin Buch, Berlin
  - Klinikum Bielefeld, Bielefeld
  - Städtisches Klinikum Dresden, Dresden
  - Universitätsklinikum TU Dresden, Dresden
  - Krankenhaus Nordwest, Frankfurt
  - Agaplesion Markus KH Frankfurt, Frankfurt am Main
  - Frankfurt Universitätsklinikum, Frankfurt am Main
  - Hamburg Onkologische Schwerpunktpraxis Eppendorf, Hamburg
  - Hämatologisch-Onkologische Praxis Altona (HOPA), Hamburg
  - Universitätsklinikum Jena, Jena
  - Ortenau Klinikum Lahr, Lahr
  - Klinikum Ludwigsburg, Ludwigsburg
  - Universitätsklinikum Lübeck, Lübeck
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Marburg, Marburg
  - Klinikum der Universität München Großhadern, München
  - Klinikum r.d. Isar, München
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Weiden, Weiden
  - Helios Dr. Horst Schmidt Kliniken, Wiesbaden
  - Klinikum Wolfsburg, Wolfsburg

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared